CLINICAL TRIAL: NCT03478007
Title: Low-Cost Tool for Compliance and Treatment-Tracking of Low Back Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Innovative Design Labs (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kenton R. Kaufman, PhD, PE, Professor of Biomedical Engineering, College of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-002177; R44AG055152-02A1 (NIH)
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Low Back Pain
Keywords: Exercise Compliance; Health Coaching
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Treatment (No Intervention): Usual standard of care (exercises)
- Intervention Technology Only (Experimental): Exercises with technology alone
  Interventions: Device: Intervention Technology
- Intervention Technology Plus Coaching (Experimental): Exercises with technology plus coaching
  Interventions: Device: Intervention Technology Plus Coaching

INTERVENTIONS:
Device: Intervention Technology — Subjects will perform their exercises using the provided monitoring device. They will be able to contact the investigators with questions regarding the use of the monitoring device, however, no encouragement or coaching will be provided
  Arms: Intervention Technology Only
Device: Intervention Technology Plus Coaching — Subjects will perform their exercises using the provided monitoring device. They will also be coached by a trained health coach through a weekly call.
  Arms: Intervention Technology Plus Coaching

SUMMARY:
The purpose of the study is to develop, design and implement an easy-to-use, cloud-enabled software for patients with low back pain and evaluate the effect of the system on compliance and quality of life. The investigators hypothesize that a device which measures compliance to physical therapy regimens in patients with low back pain will increase patient participation.

DETAILED DESCRIPTION:
Innovative Design Labs (IDL) proposes to develop and deploy a low-cost measurement system which tracks exercise compliance and enables remote health coaching for patients with low back pain. The system will consist of a series of small motion sensors built into a custom designed harness which connect wirelessly to the user's tablet or smartphone. A software application will guide the patient through the exercise routine while the sensor system monitors their motion, classifies exercise completion, and tracks their progress through the protocol. The results of the routine will be securely uploaded to caregivers where they can monitor progress, modify the patient's exercise prescription, and offer encouragement and coaching to continue the therapy. This research program aims to enable the long term treatment-tracking of patients with chronic low back pain.

ELIGIBILITY:
Inclusion

* 18 years or older
* Diagnosis of chronic low back pain (> 3 months duration)
* Have a current prescription for at-home exercises for chronic low back pain

Exclusion

* Patients with a high likelihood of being lost to follow-up or contact
* Patients with an inability to provide good data or follow commands
* Patients with an inability to do mild exercise
* Patients with a history of spine surgery that included instrumentation or hardware
* Patients who are taking opioid medication chronically without reasonable reduction in pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Change in Back Disability Related Quality of Life | Baseline and 8 weeks
  Participants will fill out the Modified Oswestry Disability Index, a 10 section questionnaire with 6 possible answers within each section. Statement 1 is graded as 0 points; statement 6 is graded as 5 points. A total score of 50 is possible and would indicate 100% disability. A score of 0-20% indicates minimal disability.

SECONDARY OUTCOMES:
Change in Overall Pain | Baseline and 8 weeks
  Participants will fill out the pain Numerical Rating Scale survey, a 4 question survey used to rate intensity of pain from a scale of 0 ("no pain") to 10 ("worst possible pain"). Pain is categorized as mile (1-3), moderate (4-6) or severe (7-10).
Degree of Compliance | 4 and 8 weeks
  Compliance collected through written diaries (control group) or electronically recorded compliance monitoring. Compliance will be defined on whether or not the subject completed the assigned exercises each day.

CONTACTS AND LOCATIONS:
Overall Officials: Kenton R Kaufman, Ph.D, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials